CLINICAL TRIAL: NCT01734967
Title: Needle-based Confocal Endomicroscopy Examination of Pancreatic Masses
Brief Title: Needle-based Confocal Endomicroscopy Examination of Pancreatic Masse
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Herlev Hospital (Other)
Responsible Party: Principal Investigator, John Gasdal Karstensen, M.D., Herlev Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: herlev
Record Dates: First submitted 2012-11-19; First posted 2012-11-28 (Estimated); Last update posted 2018-02-23 (Actual); Status verified 2018-02

CONDITIONS: Pancreatic Neoplasms; CHRONIC PANCREATITIS
Keywords: confocal laser endomicroscopy; Pancreatic Neoplasms; CHRONIC PANCREATITIS; Endoscopic ultrasound
MeSH Terms: conditions — Pancreatic Neoplasms; Pancreatitis, Chronic | interventions — Endoscopic Ultrasound-Guided Fine Needle Aspiration; Biopsy, Fine-Needle

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- needle based CLE & EUS-FNA (Experimental): The study will prospectively include patients referred to our department for EUS and EUS-FNA of suspected pancreatic masses during a 12 months period. The indication for this investigation will be based on the patient's clinical history and previous imaging studies (abdominal ultrasound, CT scan, MRI).
  Interventions: Device: needle based CLE; Procedure: EUS-FNA

INTERVENTIONS:
Device: needle based CLE — EUS-nCLE will be performed after EUS identification of the pancreatic tumor / lymph node / liver metastasis:
  The confocal microprobe will be preloaded in a 19G FNA needle as previously described and advanced into the lesion under EUS guidance.
  nCLE examination will follow after the intravenous administration of the contrast agent (2.5 ml fluorescein 10%).
  Image data will be stored digitally for offline analysis.
  Other Names: nCLE
Procedure: EUS-FNA — Endoscopic ultrasound (EUS) is an established tool in pancreatic masses used both for diagnosis, but also for staging purposes. Additionally, EUS enables guided fine needle aspiration (FNA), which is currently recommended as the first-line procedure whenever a pathological diagnosis is required.
  Other Names: Endoscopic ultrasound with fine-needle aspiration

SUMMARY:
Introduction: Pancreatic cancer is one of the most aggressive malignancies with only 5% of patients being alive at five years. EUS (endoscopic ultra sound) is an established, sensitive diagnostic tool in pancreatic cancer and for staging purposes. Additionally, EUS enables guided fine needle aspiration (FNA), which is currently recommended as the first-line procedure whenever a pathological diagnosis is required. However, EUS-FNA as a sampling method has its drawbacks, due to a relatively low negative predictive value. Confocal laser endomicroscopy has emerged in recent years as a novel method that enables in vivo microscopic analysis during ongoing endoscopy. Recently, confocal laser endomicroscopy has gone beyond the superficial luminal indications with the development of a new microprobe, i.e. a flexible laser probe (nCLE) that can pass through a 19-gauge needle. Combined with EUS, descriptive criteria for the diagnosis of pancreatic cystic neoplasm has been developed in a multicentre trial. However, only a limited number of cases of solid pancreatic masses have been described with nCLE.

Aim and Method: To describe confocal imaging criteria for pancreatic masses, lymph nodes or liver metastases identified during EUS procedures performed for pancreatic cancer staging (EUS-nCLE), while evaluating also the feasibility and safety of nCLE examination. The hypothesis is that EUS-nCLE could allow targeted tissue sampling of pancreatic lesions resulting in more accurate diagnosis. XX patients were included all presenting with a clinical suspicion of pancreatic cancer or imaging studies showing a pancreatic mass. During the procedure an nCLE preloaded 19G FNA needle was advanced into the lesion under EUS guidance. A contrast agent was administered intravenously (2.5 ml fluorescein 10%). The data was stored digitally for post procedural analysis. Afterwards EUS-FNA was performed for cytology smears to enable a final pathological diagnosis. Correlations between the nCLE images and the conventional pathology were identified.

DETAILED DESCRIPTION:
Background Pancreatic cancer is one of the most aggressive gastrointestinal malignancies with mortality rates following closely the incidence rates. The incidence is increasing and the prognosis is grim especially because of late diagnosis and metastatic potential. While surgical treatment is currently the only potential curative intervention, 80-85% of the PC cases are unfortunately detected in late unresectable stages of the disease. In spite of advances in the diagnosis and management of pancreatic cancer less than 5% of patients are alive at five years.

Endoscopic ultrasound (EUS) represents a highly valuable tool in the management of pancreatic cancer patients. As a minimally invasive technique that enables high-resolution imaging of the pancreatic parenchyma and surrounding structures it is considered the method of choice for the detection of clinically suspected pancreatic tumors, with a negative predictive value close to 100%. Its diagnostic sensitivity was shown by previous studies to be superior compared to other imaging techniques, especially in the case of smaller tumors. Additionally EUS enables guided fine needle aspiration (EUS-FNA) which is currently recommended as the firs-line procedure whenever pathological diagnosis is required. However, EUS-FNA as a sampling technique has its drawbacks, mainly represented by the relatively low negative predictive value in diagnosing pancreatic cancer. It thus cannot reliably rule out a diagnosis of malignancy and patients with high clinical suspicion usually need repeated FNA.

Confocal laser endomicroscopy has emerged in recent years as a novel technique that actually enables in vivo microscopic analysis during ongoing endoscopy. Endomicroscopy can be performed either with dedicated (eCLE) or with miniprobe-based systems (pCLE). It is a contrast based technique, the most widely used agent being the intravenously administered fluorescein. The probe-based endomicroscopy system consists of a flexible catheter probe representing a bundle of optical fibers linked to a micro-objective, a laser scanning unit and the control and acquisition software (Cellvizio; Mauna Kea Technology, Paris, France). The flexible confocal miniprobes were specifically designed to be passed through the working channels of standard endoscopes, biliary catheters or cholangioscopes and thus the pCLE system can be easily integrated in any endoscopy unit. The principle of the technique is based on a laser beam of defined wavelength being focused towards the targeted tissue and the recaptured signal is displayed as 'optical biopsies' in a single horizontal plane.

The potential role of CLE has been explored in pathology of both upper and lower gastrointestinal tract, showing good accuracy for predicting the final histopathological diagnosis based on immediate evaluation of tissue and vascular patterns. Recently CLE has gone beyond the superficial luminal indications with the development of a new microprobe, i.e. a flexible probe thin enough that it can be passed through a 19-gauge needle. Thus under EUS guidance solid organs can be accessed for real-time microscopic information. nCLE imaging of abdominal organs has been so far achieved in animal models. The feasibility of the technique was also proved in a clinical study and descriptive criteria for the diagnosis of pancreatic cystic neoplasm were developed from a multicentre trial. However, only a limited number of cases of pancreatic solid masses have been described with nCLE.

Aim The aim of the proposed study is to describe confocal imaging criteria for pancreatic masses, lymph nodes or liver metastases identified during EUS procedures performed for pancreatic cancer staging (EUS-nCLE), while evaluating also the feasibility and safety of nCLE examination. The hypothesis is that EUS-nCLE could allow targeted tissue sampling of pancreatic lesions resulting in more accurate diagnosis. With further validation of the technique real-time pathological diagnosis could be obtained with immediate initiation of the adequate therapy after a single investigation.

Patients The study will prospectively include patients referred to our department for EUS and EUS-FNA of suspected pancreatic masses during a 12 months period. The indication for this investigation will be based on the patient's clinical history and previous imaging studies (abdominal ultrasound, CT scan, MRI).

Patients will be selected according to the following criteria used throughout the study:

Data collected for each participant will include:

* Personal data (name, surname, age, sex)
* EUS variables (tumor characteristics)
* Histological and immunohistochemical findings (final diagnosis)

Imaging tests All patients with a suspicion (clinical, US, CT/MRI) of pancreatic masses will be evaluated by EUS, nCLE and EUS-FNA for pathological diagnosis.

For EUS examination linear instruments will be used to perform complete examination of the pancreas.

Tumor characteristics (echogenicity, echostructure, size, vascular invasion) will be described.

The presence of regional lymph nodes will be reported with their maximal size, echogenicity, shape and margins.

Identification of liver metastasis will also be looked upon.

EUS-nCLE will be performed after EUS identification of the pancreatic tumor / lymph node / liver metastasis:

The confocal microprobe will be preloaded in a 19G FNA needle as previously described and advanced into the lesion under EUS guidance.

nCLE examination will follow after the intravenous administration of the contrast agent (2.5 ml fluorescein 10%).

Image data will be stored digitally for offline analysis. EUS-FNA will be also performed after image acquisition for cytology smears and cell blocks to enable a final pathological diagnosis Confocal images will be analyzed during the examination by the principal investigator, with clinical and other procedural information in mind. In a second step offline analysis, the correlations between representative confocal images and classical hematoxylin and eosin sections will be identified.

Final diagnosis The final diagnosis will be based on EUS-FNA cytology and/or histological specimens in those patients that will be further referred for surgery. Pathology samples obtained from duodeno-pancreatectomies or caudal pancreatectomies done with curative intent, as well as microhistological fragments obtained through EUS-FNA biopsy will be processed by paraffin embedding with usual stainings (haematoxylin-eosin), with subsequent immune-histochemistry where necessary.

For the patients without positive cytology or histology the diagnosis will be based on EUS tumor characteristics and other relevant information (clinical, imaging tests) with follow-up for at least six months.

ELIGIBILITY:
Inclusion criteria

* Age > 18 years old, male or female
* Patients diagnosed with solid pancreatic masses with an indication for EUS-FNA
* Signed informed consent for EUS with FNA and nCLE examination

Exclusion criteria

* Failure to provide informed consent
* Patients with a contraindication for EUS-FNA
* Known allergy to fluorescein
* Pregnant or breast-feeding patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2012-11 (Actual); Primary Completion 2015-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Describe confocal imaging criteria for pancreatic masses, lymph nodes or liver metastases | 6 month
  Tumor characteristics (EUS) (echogenicity, echostructure, size, vascular invasion) will be described.
  EUS-nCLE will be performed after EUS identification of the pancreatic tumor / lymph node / liver metastasis:
  Confocal images will be analyzed to correlate representative confocal images and classical hematoxylin and eosin sections.
  The final diagnosis will be based on EUS-FNA cytology and/or histological specimens in those patients that will be further referred for surgery. For the patients without positive cytology or histology the diagnosis will be based on EUS tumor characteristics and other relevant information (clinical, imaging tests) with follow-up for at least six months
  The outcome is fully descriptive.

SECONDARY OUTCOMES:
Safety | 30 days
  Number of adverse events related til the procedure
Feasibility | 1 day
  Feasibility of nCLE examination measured by the number of patients, where nCLE is accomplished

CONTACTS AND LOCATIONS:
Overall Officials: john G Karstensen, M.D., Principal Investigator — Copenhagen University Hospital at Herlev
Locations (2):
- Copenhagen University Hospital Herlev, Herlev, Denmark
- Research Center of Gastroenterology and Hepatology,, Craiva, Romania

REFERENCES:
- [Background] Vincent A, Herman J, Schulick R, Hruban RH, Goggins M. Pancreatic cancer. Lancet. 2011 Aug 13;378(9791):607-20. doi: 10.1016/S0140-6736(10)62307-0. Epub 2011 May 26. PMID 21620466
- [Background] Sharma C, Eltawil KM, Renfrew PD, Walsh MJ, Molinari M. Advances in diagnosis, treatment and palliation of pancreatic carcinoma: 1990-2010. World J Gastroenterol. 2011 Feb 21;17(7):867-97. doi: 10.3748/wjg.v17.i7.867. PMID 21412497
- [Background] Saftoiu A, Vilmann P. Role of endoscopic ultrasound in the diagnosis and staging of pancreatic cancer. J Clin Ultrasound. 2009 Jan;37(1):1-17. doi: 10.1002/jcu.20534. PMID 18932265
- [Background] DeWitt J, Devereaux B, Chriswell M, McGreevy K, Howard T, Imperiale TF, Ciaccia D, Lane KA, Maglinte D, Kopecky K, LeBlanc J, McHenry L, Madura J, Aisen A, Cramer H, Cummings O, Sherman S. Comparison of endoscopic ultrasonography and multidetector computed tomography for detecting and staging pancreatic cancer. Ann Intern Med. 2004 Nov 16;141(10):753-63. doi: 10.7326/0003-4819-141-10-200411160-00006. PMID 15545675
- [Background] Iglesias Garcia JJ, Larino Noia J, Alvarez Castro A, Cigarran B, Dominguez Munoz JE. Second-generation endoscopic ultrasound elastography in the differential diagnosis of solid pancreatic masses. Pancreatic cancer vs. inflammatory mass in chronic pancreatitis. Rev Esp Enferm Dig. 2009 Oct;101(10):723-30. doi: 10.4321/s1130-01082009001000009. English, Spanish. PMID 19899942
- [Background] Dumonceau JM, Polkowski M, Larghi A, Vilmann P, Giovannini M, Frossard JL, Heresbach D, Pujol B, Fernandez-Esparrach G, Vazquez-Sequeiros E, Gines A; European Society of Gastrointestinal Endoscopy. Indications, results, and clinical impact of endoscopic ultrasound (EUS)-guided sampling in gastroenterology: European Society of Gastrointestinal Endoscopy (ESGE) Clinical Guideline. Endoscopy. 2011 Oct;43(10):897-912. doi: 10.1055/s-0030-1256754. Epub 2011 Aug 12. PMID 21842456
- [Background] Becker V, Wallace MB, Fockens P, von Delius S, Woodward TA, Raimondo M, Voermans RP, Meining A. Needle-based confocal endomicroscopy for in vivo histology of intra-abdominal organs: first results in a porcine model (with videos). Gastrointest Endosc. 2010 Jun;71(7):1260-6. doi: 10.1016/j.gie.2010.01.010. Epub 2010 Apr 24. PMID 20421104
- [Background] Konda VJ, Aslanian HR, Wallace MB, Siddiqui UD, Hart J, Waxman I. First assessment of needle-based confocal laser endomicroscopy during EUS-FNA procedures of the pancreas (with videos). Gastrointest Endosc. 2011 Nov;74(5):1049-60. doi: 10.1016/j.gie.2011.07.018. Epub 2011 Sep 15. PMID 21924718
- [Derived] Karstensen JG, Cartana T, Klausen PH, Hassan H, Popescu CF, Saftoiu A, Vilmann P. Endoscopic ultrasound-guided needle-based confocal laser endomicroscopy: a pilot study for use in focal pancreatic masses. Pancreas. 2015 Jul;44(5):833-5. doi: 10.1097/MPA.0000000000000345. No abstract available. PMID 26061561